CLINICAL TRIAL: NCT06906705
Title: High Frequency Ultrasound Imaging for Intraoperative Lymph Nodal Assessment in Gynecological Cancer: From Image-guided Surgery to Radiomics Applications
Brief Title: High-frequency Ultrasound for Intraoperative Lymph Node Assessment in Gynecological Cancer: From Surgery to Radiomics
Acronym: RHINOCERUS
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Canon Medical Systems Europe B.V (Unknown)
Responsible Party: Sponsor
Other Study IDs: 7480
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-03

CONDITIONS: Gynecologic Cancer
Keywords: ovarian cancer; endometrial cancer; cervical cancer; vulvar cancer; HFUS
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lymph node assessment is crucial in gynecological cancers (ovarian, endometrial, cervical, and vulvar), as nodal involvement significantly impacts prognosis and treatment. Despite high morbidity, systematic lymphadenectomy has been widely used for staging and treatment planning. However, in most cases, lymph nodes are free from metastasis, making the procedure unnecessary and exposing patients to severe complications such as lymphedema and infections.

Sentinel lymph node (SLN) evaluation has emerged as a less invasive alternative, reducing unnecessary lymphadenectomies. However, SLN techniques face challenges, including detection failures, inaccurate frozen section analysis, and imaging limitations like false negatives in FDG PET/CT scans. The need for improved intraoperative imaging techniques is emphasized to enhance lymph node assessment, minimize surgical risks, and better tailor treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing surgery for gynecological malignancies (ovarian, endometrial, cervical, and vulvar cancer)
* Need for nodal excision (staging or cytoreductive reasons)
* 18-99 years old
* Absence of contemporary lymphatic diseases
* Absence of previous oncological disease in the last 5 years
* Willingness to participate in the study and to provide informed consent

Exclusion Criteria:

* Previous radiotherapy treatments
* Previous chemotherapy treatments

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Gynecology Oncology Unit in Fondazione Policlinico A. Gemelli
  IRCCS, Italy, Rome with a diagnosis of gynecological malignancy requiring surgical lymph nodes harvest will be evaluated for the enrolment.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of HFUS Accuracy in Detecting Lymph Node Metastases in Gynecological Cancer | Days 20
  The aim of this prospective trial is to report the sensivity, specificity, NPV, PPV and accuracy of HFUS in the metastasis detection (macro, micro and ITCs) from fresh, unstained ex vivo/in vivo lymph node samples.

SECONDARY OUTCOMES:
Minimum Size Detection Limit of HFUS Imaging | 2 minutes
  To assess the lowest size detectable with the adopted imaging technique
Development of a Radiomic Algorithm for Lymph Node Assessment | 6 months
  To develop a radiomic algorithm for the assesment of the lymphn node status

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Carla Testa, Professor, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy